CLINICAL TRIAL: NCT03257826
Title: The Effect of Percutaneous Kirschner Wire Technique in Management of Congenital Pseudarthrosis of Tibia Under One Year Old
Brief Title: The Effect of Percutaneous Kirschner Wire Technique in Management of CPT Under One Year Old
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hunan Children's Hospital (Other Government)
Collaborators: Guangzhou Women and Children's Medical Center (Other); Shenzhen Children's Hospital (Other Government); Tongji Hospital (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Wuhan Women and Children's Medical Center (Other); Foshan Hospital of Traditional Chinese Medicine (Other); Dalian Children's Hospital (Other); Children's Hospital of Chongqing Medical University (Other); Kunming Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HN04
Record Dates: First submitted 2017-08-15; First posted 2017-08-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Congenital Pseudarthrosis of Tibia
Keywords: congenital pseudarthrosis of the tibia; age of surgery; Percutaneous Kirschner wire
MeSH Terms: interventions — Bone Wires

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- surgery (Experimental): Percutaneous Kirschner wire
  Interventions: Device: kirschner wire

INTERVENTIONS:
Device: kirschner wire — retrograde percutaneous kirschner wire was applied to stabilize the tibia.

SUMMARY:
The aim of this study was to investigate the effect of percutaneous kirschner wire in management of Congenital Pseudarthrosis of Tibia in children younger than 1 year of age. This study was to determine the union rates of congenital pseudarthrosis in children operated before 1 year of age to identify growth abnormalities in the affected limb ,including ankle valgus,tibia valgus,and shortening.

DETAILED DESCRIPTION:
Currently, the timing of surgery for congenital pseudarthrosis of the tibia is a controversial issue. The investigators use percutaneous kirschner wire technique to manage the Congenital Pseudarthrosis of Tibia in children younger than 1 year of age.To investigate the effect of percutaneous kirschner wire in management of Congenital Pseudarthrosis of Tibia in children younger than 1 year of age. Bone uion rate,average time of healing, ankle valgus, limb length discrepancy, tibia axis alignment are recorded and evaluated.

ELIGIBILITY:
Inclusion Criteria:

* All patients did not undergo procedures
* Patients with Crawford type IV CPT treated with Percutaneous Kirschner wire techniques
* The age during surgery was less than 12 months old

Exclusion Criteria:

* Patients with pseudarthrosis of tibia caused by trauma,infection, etc

Ages: 1 Month to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2015-08-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Primary union score (range,4-12 score) | 9 months post-operation
  X ray score from tibia pseudarthrosis in anterior and posterior (AP )and lateral X ray. ("RUST" score:radiographic union scoring system for tibial fracture healing)

SECONDARY OUTCOMES:
Refracture（Cortical discontinuity) | 0.5 , 1,2,3,4,5,6,7,8,9,10 years after the fracture is healed
  Refracture was defined as an obvious fracture（Cortical discontinuity) on a plain radiograph,following the union at the site of the tibia.
Residual Deformity-proximal tibia angulation(range,0°-90°) | pre-operation and 0.5 , 1,2,3,4,5,6,7,8,9,10 years post-operation ]
  measurement of the angulation of proximal tibia in anterior and posterior (AP )and lateral X ray.Proximal tibial valgus is created by the intersection of a line parallel to the proximal physis and another line along the axis of the proximal third of diaphysis in the tibia.
Residual Deformity-Limb length discrepancy | pre-operation and 0.5 , 1,2,3,4,5,6,7,8,9,10 years post-operation
  measurement of the length difference of both tibia in AP and lateral X ray.Picture Archiving and Communication System (PACS) is used to measure the length of the tibia (The investigators measure the distance between the midpoint of the proximal tibial epiphyseal plate and the midpoint of distal tibia epiphyseal plate).
Residual Deformity-ankle valgus angulation(range,0°-90°) | pre-operation and 0.5 , 1,2,3,4,5,6,7,8,9,10 years post-operation
  measurement of the angulation between the distal tibia and ankle joint.Ankle valgus is assessed by the tibiotalar angle measured at the intersection of the mid-diaphyseal line of the tibia and a line drawn across the flat subchondral line of the talar dome.

CONTACTS AND LOCATIONS:
Overall Officials: Haibo Mei, MD, Study Director — Hunan Children's Hospital
Locations (1):
- Kun Liu, Changsha, Hunan, China